CLINICAL TRIAL: NCT07287904
Title: A Retrospective Analysis Study on Predicting the Efficacy of Targeted Therapy in Lung Cancer Patients With EGFR Mutations Based on AI-driven Multimodal Data
Brief Title: Prediction of Targeted Therapy Efficacy in EGFR-mutant Lung Cancer Patients Using AI-based Multimodal Data
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: AIEF20250825
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer (NSCLC); EGFR Activating Mutation; Adenocarcinoma Lung; Postoperative Adjuvant Therapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comprehensive analysis through laboratory tests, imaging techniques, and clinical data — Extract radiomics features of the tumor and peritumoral regions from preoperative CT images, H&E-stained digital pathology whole-slide images, and genetic test reports, and integrate them with multidimensional pathological features and gene expression distribution characteristics to construct a radiopathogenomic multi-omics modality, providing more precise prognostic assessment for targeted therapy in lung cancer patients.

SUMMARY:
The main purpose of this study is to explore the value of multimodal imaging information and models in predicting the prognosis of EGFR-positive non-small cell lung cancer patients undergoing targeted therapy, providing a basis for selecting suitable populations for precise tumor treatment and corresponding therapy. We retrospectively analyzed patient case data, extracted preoperative CT images, H&E-stained whole-slide digital pathology images, and pre- or postoperative genetic testing reports to extract radiomic features of tumor and peritumoral regions. These features were combined with multidimensional pathological features and gene expression distribution characteristics to construct a multimodal radiopathogenomic model, offering more precise prognostic evaluation for lung cancer patients receiving targeted therapy.

DETAILED DESCRIPTION:
This study is an observational study, aiming to retrospectively include data from 500 patients diagnosed with stage IB-IIIA invasive lung adenocarcinoma who underwent radical surgery at Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, from January 2021 to December 2024, along with data from a total of 1,000 patients from other multi-center sites. The study will collect and record information on subjects' demographics, pathology, imaging, genetic testing, and clinical characteristics via the hospital's electronic medical record system. Patient survival status will be obtained through telephone follow-ups and home visits. Radiomic features of the tumor and peritumoral regions will be extracted from preoperative CT images, H&E-stained digital whole-slide pathology images, and genetic testing reports. These will be combined with multi-dimensional pathological features and gene expression distribution characteristics from the patient cases to construct a multi-omics model integrating imaging, pathology, demographics, and genetics, providing a more precise prognostic assessment for targeted therapy in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, undergoing radical surgery for lung cancer (R0 resection);
2. Postoperative pathological stage IB-IIIA, pathology confirmed as adenocarcinoma;
3. EGFR gene testing positive, EGFR 19del/L858R mutation;
4. Receiving postoperative EGFR-TKI targeted adjuvant therapy;
5. Complete and clear preoperative imaging data, genetic testing report, and pathology report available.

Exclusion Criteria:

1. Patients negative for EGFR;
2. Incomplete surgical resection (R1, R2);
3. Did not receive EGFR-TKI targeted therapy after surgery;
4. Recurrent or advanced stage patients;
5. Incomplete preoperative or postoperative data;
6. Patients who died within 30 days post-surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospectively included data from 1000 patients diagnosed with stage IB-IIIA invasive lung adenocarcinoma with EGFR mutations who underwent radical surgery from January 2021 to December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
DFS | two years
  The endpoint of this study was disease-free survival (DFS), defined as the time interval from surgery to the first recurrence or death,assessed up to 24 months。

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Dong, Dr, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vaidya P, Bera K, Gupta A, Wang X, Corredor G, Fu P, Beig N, Prasanna P, Patil PD, Velu PD, Rajiah P, Gilkeson R, Feldman MD, Choi H, Velcheti V, Madabhushi A. CT derived radiomic score for predicting the added benefit of adjuvant chemotherapy following surgery in stage I, II resectable non-small cell lung cancer: a retrospective multicohort study for outcome prediction. Lancet Digit Health. 2020 Mar;2(3):e116-e128. doi: 10.1016/S2589-7500(20)30002-9. Epub 2020 Feb 13. PMID 33334576
- [Result] Chen M, Lu H, Copley SJ, Han Y, Logan A, Viola P, Cortellini A, Pinato DJ, Power D, Aboagye EO. A Novel Radiogenomics Biomarker for Predicting Treatment Response and Pneumotoxicity From Programmed Cell Death Protein or Ligand-1 Inhibition Immunotherapy in NSCLC. J Thorac Oncol. 2023 Jun;18(6):718-730. doi: 10.1016/j.jtho.2023.01.089. Epub 2023 Feb 10. PMID 36773776
- [Result] Lin H, Hua J, Gong Z, Chen M, Qiu B, Wu Y, He W, Wang Y, Feng Z, Liang Y, Long W, Li R, Kuang Q, Chen Y, Lu J, Luo S, Zhao W, Yan L, Chen X, Shi Z, Xu Z, Mo Z, Liu E, Han C, Cui Y, Yang X, Chen X, Liu J, Pan X, Madabhushi A, Lu C, Liu Z. Multimodal radiopathological integration for prognosis and prediction of adjuvant chemotherapy benefit in resectable lung adenocarcinoma: A multicentre study. Cancer Lett. 2025 Apr 28;616:217557. doi: 10.1016/j.canlet.2025.217557. Epub 2025 Feb 13. PMID 39954935